CLINICAL TRIAL: NCT02288494
Title: Acid Base Balance of ICU Patients With Severe Hypoalbuminemia, Before and After an Albumin Infusion, Using Stewart Approach
Acronym: STEWALB
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0204
Record Dates: First submitted 2014-09-12; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Hypoalbuminemia; Adult ICU Patient; Stewart Approach for Acid Base Disorders; Human Albumin Perfusion
Keywords: hypoalbuminemia; -acid base balance; acid base disorders; critical ill; Stewart approach; human albumin infusion
MeSH Terms: conditions — Hypoalbuminemia

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- hypoalbuminemia: The primary purpose was to describe the acid base balance of ICU patients with severe hypoalbuminemia using Stewart's approach for acid base disorders, before and after an human albumin perfusion
  Interventions: Other: stewart approach

INTERVENTIONS:
Other: stewart approach — Prospective study, for ICU patient with severe hypoalbuminemia < 20g/L, determining biological parameters from Stewart approach for acid base disorders (pH, SIDe, SIDa, SIG, Atot, PaCO2) before, and at 1hour, 2hours and 24 hours after a 200mL 20% human al Clinical parameters (respiratory, haemodynamic, neurologic) were also collected at the same times.

SUMMARY:
The primary purpose was to describe the acid base balance of ICU patients with severe hypoalbuminemia using Stewart's approach for acid base disorders, before and after an human albumin perfusion.

DETAILED DESCRIPTION:
Prospective study, for ICU patient with severe hypoalbuminemia < 20g/L, determining biological parameters from Stewart approach for acid base disorders (pH, SIDe, SIDa, SIG, Atot, PaCO2) before, and at 1hour, 2hours and 24 hours after a 200mL 20% human albumin perfusion (the consensus conference ANAES of 1995 recommands to correct hypoalbuminemia below 20g/L).

Clinical parameters (respiratory, haemodynamic, neurologic) were also collected at the same times.

ELIGIBILITY:
Inclusion Criteria:

* serum albuminemia < 20g/L
* adult ICU patient
* Arterial line

Exclusion Criteria:

* albumin allergy
* pregnancy
* congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with severe hypoalbuminemia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
changes in pH and independent pH determinants using Stewart approach | at 1 hour, 2 hours and 24 hours after a 200mL of 20% human albumin perfusion.

SECONDARY OUTCOMES:
changes in neurologic parameters | at 1 hour, 2 hours and 24 hours after a 200mL of 20% human albumin perfusion.
changes in hemodynamic parameters | at 1 hour, 2 hours and 24 hours after a 200mL of 20% human albumin perfusion.
changes in respiratory parameters | at 1 hour, 2 hours and 24 hours after a 200mL of 20% human albumin perfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Julien PASCAL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France